CLINICAL TRIAL: NCT05484453
Title: Validation of the Eye Screeningtest GoCheckKids (GCK) for the Detection of Amblyopia Risk Factors in Toddlers in Flanders.
Brief Title: Validation of the GoCheck Kids® Eye Screeningtest in Infants in Flanders
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64113
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Amblyopia; Infant
Keywords: Eye screening
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GoCheckKids screening: GoCheckKids screening at the Child And Family Agency at the age of 12-15 months (+- 1 month) are invited to undergo a complete eye examination by an ophthalmologist for evaluation of amblyopia risk factors.
  Interventions: Diagnostic Test: Complete Eye Examination by Ophthalmologist

INTERVENTIONS:
Diagnostic Test: Complete Eye Examination by Ophthalmologist — complete eye examination (gold standard) including cover test, biomicroscopy and cycloplegic refraction with retinoscopy, performed by an ophthalmologist.

SUMMARY:
The aim is to validate the new GoCheck Kids application as automatic eye screener for preschool children (<3 years of age) at 'Child and Family' agency. Sensitivity, specificity, positive and negative predictive value of the GoCheck Kids screening tool are the endpoints of this study.

DETAILED DESCRIPTION:
Comparison of the results of the GoCheck Kids application on iPhone with a complete eye examination (gold standard) including cycloplegic refraction with retinoscopy, performed by an ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* GoCheck Kids (GCK) evaluation at Child and Family Agency at the age between 11-16 months.

Exclusion Criteria:

* Allergy for the used cycloplegia cyclopentolate 0.5%.
* Any history of ocular surgery
* The time window between GCK measurement and the complete eye examination may not exceed 2 months.
* The parents or legal representatives of the child do not understand or speak Dutch, French or English.

Ages: 11 Months to 16 Months | Sex: All
Age Groups: Child
Study Population: Children who undergo GCK evaluation at the Child And Family Agency consultation
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Day 1
  Sensitivity of GCK eye screener
Specificity | Day 1
  Specificity of GCK eye screener
Positive predictive value | Day 1
  Positive predictive value of GCK eye screener
Negative predictive value | Day 1
  Negative predictive value of GCK eye screener

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cassiman, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No